CLINICAL TRIAL: NCT04246684
Title: Short-course Radiotherapy Versus Chemoradiotherapy, Followed by Consolidation Chemotherapy, and Selective Organ Preservation for MRI-defined Intermediate and High-risk Rectal Cancer Patients
Brief Title: Short RT Versus RCT,Followed by Chemo.and Organ Preservation for Interm and High-risk Rectal Cancer Patients
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Prof. Dr. med. Claus Rödel (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Claus Rödel, Prof. Dr. med., Goethe University
Organization: Goethe University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACO/ARO/AIO-18.1
Record Dates: First submitted 2020-01-23; First posted 2020-01-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Rectal Cancer Stage III
MeSH Terms: conditions — Rectal Neoplasms | interventions — Oxaliplatin; Fluorouracil; Leucovorin; Capecitabine

STUDY DESIGN:
Intervention Model Description: Investigator-driven
Who Masked: Investigator
Masking Description: multicentre, open-labeled, Phase III study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Active Comparator): In the control arm patients receive 5x5 Gy followed by 9 cycles of consolidation chemotherapy mFOLFOX6 or alternatively 6 cycles of CAPOX, followed by re-staging at week 22-24 as established as new preferred neoadjuvant regimen by the RAPIDO trial.
  Interventions: Drug: Oxaliplatin, 85 mg/m2; Drug: 5FU; 2400 mg/m2; Drug: Folinic Acid, 400 mg/m2; Radiation: Radiotherapy control, 5x5 Gy: 25 Gy; Drug: Capecitabine, 1000 mg/m2; Drug: Oxaliplatin, 130 mg/m2
- Experimental arm (Experimental): The experimental arm starts with Fluoropyrimidin/Oxaliplatin-based CRT (1.8 Gy to 45 Gy to the primary tumor and pelvic lymph nodes; followed by sequential boost of 9 Gy to the gross tumor volume) followed by consolidation chemotherapy with 6 cycles mFOLFOX6 or alternatively 4 cycles CAPOX, followed by re-staging at week 22-24. In both arms, for patients achieving a clinical complete response (cCR), as strictly assessed by clinical investigation, endoscopy and MRI, a W&W option with close follow-up is scheduled. In case of non-complete response, immediate TME surgery is performed.
  Interventions: Drug: 5FU, 250 mg/m2; Drug: 5FU, 2400 mg/m2; Drug: Oxaliplatin 50 mg/m2; Drug: Folinic Acid, 400 mg/m2; Drug: Capecitabine, 1000 mg/m2; Drug: Oxaliplatin 85 mg/m2; Radiation: radiotherapy experimental, 30 x 1,8 Gy: 54 Gy; Drug: Capecitabine, 825 mg/m2; Drug: Oxaliplatin, 130 mg/m2

INTERVENTIONS:
Drug: Oxaliplatin, 85 mg/m2 — 85 mg/m2,2h-civ, day 22, 36, 50, 64, 78, 92, 106, 120, and 134 of therapy
  Other Names: Control arm
  Arms: Control arm
Drug: 5FU; 2400 mg/m2 — 2400 mg/m2, 46h-civ, day 22, 36, 50, 64, 78, 92, 106, 120, 134 of therapy for Control arm
  Other Names: 5-FU, control arm
  Arms: Control arm
Drug: 5FU, 250 mg/m2 — 250 mg/m2 per day, civ, on day 1-14, day 22-35 of radiotherapy;
  Other Names: Experimental arm: 5-FU
  Arms: Experimental arm
Drug: 5FU, 2400 mg/m2 — 2400 mg/m2,46h-civ, d64, d78, d92, d106, d120, d134 of therapy
  Other Names: experimental arm
  Arms: Experimental arm
Drug: Oxaliplatin 50 mg/m2 — 50 mg/m2, 2h-civ, d1, d8, d21, d29 of radiotherapy and
  Other Names: Experimental arm
  Arms: Experimental arm
Drug: Folinic Acid, 400 mg/m2 — 2h-civ day 22, 36, 50, 64, 78, 92, 106, 120, and 134 of therapyfor Control arm; 400 mg/m2, 2h-civ d 64, d78, d92, d106, d120, d134 of therapy for experimental arm
  Other Names: Folinic Acid
Radiation: Radiotherapy control, 5x5 Gy: 25 Gy — Control arm: 5x5 Gy (total: 25 Gy) 5 fractions
  Arms: Control arm
Drug: Capecitabine, 1000 mg/m2 — 1000 mg/m2 (twice daily) day1-14 every three weeks instead of 5FU optional
  Other Names: Capecitabine
Drug: Oxaliplatin 85 mg/m2 — 85 mg/m2, 2h-civ, d64, d78, d92, d106, d120, d134 of therapy
  Other Names: experimental arm
  Arms: Experimental arm
Radiation: radiotherapy experimental, 30 x 1,8 Gy: 54 Gy — 30 x 1.8 Gy (total: 54 Gy), 5 fractions per week
  Arms: Experimental arm
Drug: Capecitabine, 825 mg/m2 — 825 mg/m2 bid, per os, on day 1-14, 22-35 of RT instead of 5FU optional
  Other Names: Capecitabine
  Arms: Experimental arm
Drug: Oxaliplatin, 130 mg/m2 — day1every three weeks (optional)
  Other Names: Oxaliplatin

SUMMARY:
The hereby proposed ACO/ARO/AIO-18.1 randomized trial aims to directly compare the newly established TNT concepts applying either short-course RT according to RAPIDO, or CRT according to CAO/ARO/AIO-04/-12, both followed by consolidation chemotherapy, and surgery or a watch&wait (W&W) approach for patients with clinical complete response (cCR).

The ACO/ARO/AIO-18.1 study incorporates several novel and innovative aspects to further optimize multimodal rectal cancer treatment, partly established by our preceding CAO/ARO/AIO-04 and CAO/ARO/AIO-12 randomized trials: (1) patient selection is based on strict, quality controlled MRI features of intermediate and high-risk characteristics (and, thus, complementary to our ACO/ARO/AIO-18.2 trial in "low-risk" rectal cancer), (2) the CRT regimens incorporates 5-FU/oxaliplatin with doses and intensities shown to be effective and well-tolerated without compromising treatment compliance in CAO/ARO/AIO-04, (3) the sequence of CRT, CT, and surgery/W&W adopts the TNT approach as established by our CAO/ARO/AIO-12 and OPRA trial, (4) surgical stratification allows for W&W management for strictly selected patients with clinical complete response (cCR). Thus, we hypothesize that TNT with 5-FU/oxaliplatin-CRT followed by consolidation chemotherapy may increase organ preservation while maintaining DFS as compared to RAPIDO-like short-course RT followed by consolidation chemotherapy.

DETAILED DESCRIPTION:
The primary endpoint of this trial, organ preservation, is defined as follows: survival with rectum intact, no major surgery, no stoma. Accordingly, the primary endpoint, organ preservation, will not be reached if any of the following occurs: (1) death, (2) any major surgery other than local excision (R0) performed after randomization, during TNT, at re-staging scheduled 22-24 weeks after start of TNT due to clinical non-cCR, or for any locoregional regrowth after initial cCR requiring salvage-TME, (3) any locoregional regrowth not amenable to salvage surgery, or (4) any stoma (non-re-converted protective stoma within 6 months after completion of TNT, or any stoma needed for toxicity or poor function), whichever occurs first. We hypothesized that the 3-year organ preservation rate will improve from 30% in the control arm to 40% in the investigational arm (hazard ratio of 0.76). With a power of 90% and a two-sided type I error of 5%, the sample size required to obtain a statistically significant difference is 702 patients (564 events) in total.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of rectal adenocarcinoma localised 0 - 12 cm from the anocutaneous line as measured by rigid rectoscopy (i.e. lower and middle third of the rectum)
* Staging requirements: High-resolution, thin-sliced (i.e. 3mm) magnetic resonance imaging (MRI) of the pelvis is the mandatory local staging procedure.
* MRI-defined inclusion criteria: presence of at least one of the following high-risk conditions:
* any cT3 if the distal extent of the tumor is < 6 cm from the anocutaneous line, or
* cT3c/d in the middle third of the rectum (≥ 6-12 cm) with MRI evidence of extramural tumor spread into the mesorectal fat of more than 5 mm (>cT3b), or
* cT3 with clear cN+ based on strict MRI-criteria
* cT4 tumors, or
* Tany middle/low third of rectum with clear MRI criteria for N+
* mrCRM+ (< 1mm), or
* Extramural venous invasion (EMVI+)
* Trans-rectal endoscopic ultrasound (EUS) is additionally used when MRI is not definitive to exclude early cT1/T2 disease in the lower third of the rectum or early cT3a/b tumors in the middle third of the rectum.
* Spiral-CT of the abdomen and chest to exclude distant metastases.
* Aged at least 18 years. No upper age limit.
* WHO/ECOG Performance Status 0-1
* Adequate haematological, hepatic, renal and metabolic function parameters:
* Leukocytes ≥ 3.000/mm^3, ANC ≥ 1.500/mm^3, platelets ≥ 100.000/mm^3, Hb > 9 g/dl
* Serum creatinine ≤ 1.5 x upper limit of normal
* Bilirubin ≤ 2.0 mg/dl, SGOT-SGPT, and AP ≤ 3 x upper limit of normal • Informed consent of the patient

Exclusion Criteria:

* Lower border of the tumor localised more than 12 cm from the anocutaneous line as measured by rigid rectoscopy
* Distant metastases (to be excluded by CT scan of the thorax and abdomen)
* Prior antineoplastic therapy for rectal cancer
* Prior radiotherapy of the pelvic region
* Major surgery within the last 4 weeks prior to inclusion
* Subject pregnant or breast feeding, or planning to become pregnant within 6 months after the end of treatment.
* Subject (male or female) is not willing to use highly effective methods of Contraception during treatment and for 6 months after the end of treatment.
* On-treatment participation in a clinical study in the period 30 days prior to inclusion
* Previous or current drug abuse
* Other concomitant antineoplastic therapy
* Serious concurrent diseases, including neurologic or psychiatric disorders (incl. dementia and uncontrolled seizures), active, uncontrolled infections, active, disseminated coagulation disorder
* Clinically significant cardiovascular disease in (incl. myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) < 6 months before enrolment
* Prior or concurrent malignancy < 3 years prior to enrolment in study (Exception: non-melanoma Skin cancer or cervical carcinoma FIGO stage 0-1), if the patient is continuously disease-free
* Known allergic reactions on study medication
* Known dihydropyrimidine dehydrogenase deficiency
* Psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule (these conditions should be discussed with the patient before registration in the trial).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male and female patients with histologically confirmed diagnosis of rectal adenocarcinoma localised 0 - 12 cm from the anocutaneous line as measured by rigid rectoscopy
Enrollment: 702 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2028-09-15 (Estimated)

PRIMARY OUTCOMES:
organ preservation | 3 years
  it is defined as follows: survival with rectum intact, no major surgery, no stoma. Accordingly, the primary endpoint, organ preservation, will not be reached if any of the following occurs: (1) death, (2) any major surgery other than local excision (R0) performed after randomization, during TNT, at re-staging scheduled 22-24 weeks after start of TNT due to clinical non-cCR, or for any locoregional regrowth after initial cCR requiring salvage-TME, (3) any locoregional regrowth not amenable to salvage surgery, or (4) any stoma (non-re-converted protective stoma within 6 months after completion of TNT, or any stoma needed for toxicity or poor function), whichever occurs first.

SECONDARY OUTCOMES:
Disease-free survival | 3 years
  Disease-free survival
Rate of clinical complete response after TNT: | 3 years
  TNT total neoadjuvant therapy
Rate of immediate TME after TNT | 3 years
  TNT total neoadjuvant therapy TME total mesorectal excision
Cumulative incidence of locoregional regrowth after cCR | 3 years
  cCR clinical complete response
Rate of salvage surgery (LE/TME with or APR/stoma) after locoregional regrowth APR/stoma) after locoregional regrowth | 3 years
  LE local Exision; TME: Transanale endoscopic Mikrochirurgie; APR Abdomino perineal Rectum exstirpation
Cumulative incidence of local recurrence after (salvage) surgery surgery | 3 years
  Cumulative incidence of local recurrence after (salvage) surgery
Postoperative complications of (salvage) surgery | 3 years
  Postoperative complications of (salvage) surgery
Rate of sphincter-sparing (salvage) surgery | 3 years
  Rate of sphincter-sparing (salvage) surgery
Pathological TNM-staging | 3 years
  Pathological tumor evaluations;TNM tumor staging
R0 resection rate; negative circumferential resection rate | 3 years
  R0 Removal of the tumor in healthy tissue
Tumor regression grading according to Dworak | 3 years
  pathological response from scale 1-4 poor to very good ascending
Neoadjuvant rectal score | 3 years
  Neoadjuvant rectal score from low to high values means good to poor
Quality of TME according to MERCURY | 3 years
  Tumor response using MRI scale 1-5 from good to poor descending
Acute and late toxicity assessment according to NCI CTCAE V.5.0) CTCAE V.5.0) | 3 Yeears
  CTCAE V.5.0
Quality of life C30 based on treatment arm and surgical procedures/organ preservation | 3 years
  Quality of life based on EORTC-QLQs-C30
functional outcome based on treatment arm and surgical procedures/organ preservation | 3 years
  functional outcome based on Wexner score
Quality of life CR29 based on treatment arm and surgical procedures/organ preservation | 3 years
  Quality of life based on EORTC-QLQs-CR29
Quality of life CPIN 20 based on treatment arm and surgical procedures/organ preservation | 3 years
  Quality of life based on EORTC-QLQs-CPIN20 Quality of life based on EORTC-QLQs-CPIN20
Cumulative incidence of distant metastases | 3 Years
  Cumulative incidence of distant metastases
Overall survival | 3 years
  Overall survival
Translational / biomarker studies | 3 years
  The translational research program will include proteomics, genomics and immune profile assessment in primary tumor samples as well as peripheral bloods samples (liquid biopsy).
  Tumor tissue samples and blood will be collected, processed and stored using protocols.
  Primary tumor tissue with either fresh tissue or formalin-fixed, paraffin-embedded (FFPE) tissue will be collected at two different time points: i) preoperative biopsy; ii) before/during surgical resection. Peripheral blood samples will be stored at three different time points: i) immediately before initiation of preoperative treatment (day 1); ii) during therapy assessment at week 22-24 and iii) at the time point of the first follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Claus Roedel, Prof. Dr., Study Director — clinic for radiotherapy
Locations (76):
- Germany (76):
  - Clincal Center Esslingen, Esslingen am Neckar, Baden-Wurttemberg
  - University Clinic Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - University Clinic Mannheim, Mannheim, Baden-Wurttemberg
  - Clinic Ostlab, Staufenclinic Schwaeb.Gmuend, Mutlangen, Mutlangen, Baden-Wurttemberg
  - Pi.Tri-Studien GmbH, Offenburg, Offenburg, Baden-Wurttemberg
  - Medius Clincal Center Ostfildern-Ruit, Ostfildern, Baden-Wurttemberg
  - Clinic Stuttgart, Stuttgart, Baden-Wurttemberg
  - University Clinic for Radioncology Tübingen, Tübingen, Baden-Wurttemberg
  - University Clinic Ulm, Ulm, Baden-Wurttemberg
  - Clincal Center "St. Marien" Amberg, Amberg, Bavaria
  - Clinic Bayreuth GmbH, Bayreuth, Bavaria
  - Clinical Center Coburg, Coburg, Bavaria
  - University Clinic Erlangen, Erlangen, Bavaria
  - Klinikverbund Allgäu, Kempten (Allgäu), Bavaria
  - Technical University Clinic Munich, München, Bavaria
  - Technical University Munich, München, Bavaria
  - Clincal Center "Bogenhausen" Munich, München, Bavaria
  - Hospital "Barmherzige Brüder" Regensburg, Regensburg, Bavaria
  - University Clinic Regensburg, Regensburg, Bavaria
  - Clinic Nordoberpfalz AG, Clinic Weiden, Weiden, Bavaria
  - University Clinic Würzburg, Würzburg, Bavaria
  - Clincal Center Helios Bad Saarrow, Bad Saarow, Brandenburg
  - Clincal Center Darmstadt, Darmstadt, Hesse
  - Clinic North West gGmbH Frankfurt, Frankfurt am Main, Hesse
  - Clinic Fulda, Fulda, Hesse
  - DRK Clincal Centers North Hessen Kassel, Kassel, Hesse
  - University Clinic Marburg, Marburg, Hesse
  - Sana Clinical Center Offenbach, Offenbach, Hesse
  - Lahn-Dill Clinics Wetzlar, Wetzlar, Hesse
  - MVZ Oncological Cooperation Harz, Goslar, Lower Saxony
  - University Clinic Göttingen, Göttingen, Lower Saxony
  - Hematological-Oncological Practice Dr. Oleg Rubanov, Hameln, Hamelin, Lower Saxony
  - Medical Project Hannover, Hanover, Lower Saxony
  - "St. Bernward" Clincal Center Hildesheim, Hildesheim, Lower Saxony
  - Oncology in Medicinum Hildesheim, Hildesheim, Lower Saxony
  - Oncology UnterEms, Leer, Leer, Lower Saxony
  - Pius Hospital, Oldenburg, Oldenburg, Lower Saxony
  - University Clinic Oldenburg, Oldenburg, Lower Saxony
  - Clinic Wolfsburg, Wolfsburg, Lower Saxony
  - University Clinic Rostock, Rostock, Mecklenburg-Vorpommern
  - Franziskus Hospital Bielefeld, Bielefeld, North Rhine-Westphalia
  - St. Josef Hospital of the catholic clinic Bochum, Bochum, North Rhine-Westphalia
  - Hospital Bochum, Bochum, North Rhine-Westphalia
  - Clinic Lippe GmbH (Lemgo/Detmold), Detmold, North Rhine-Westphalia
  - University Clinic Essen, Essen, North Rhine-Westphalia
  - Clinical Center "Essen Mitte", Essen, North Rhine-Westphalia
  - Clinic Maria Hilf GmbH, Mönchengladbach, North Rhine-Westphalia
  - Brother clinic St. Josef, Paderborn, Paderborn, North Rhine-Westphalia
  - St. Vincenz Hospital Paderborn, Paderborn, North Rhine-Westphalia
  - Prosper Hospital Recklinghausen, Recklinghausen, North Rhine-Westphalia
  - Mathias-Spital, Rheine, Rheine, North Rhine-Westphalia
  - Evangelical Clinic Wesel, Wesel, North Rhine-Westphalia
  - University Clinic Mainz, Mainz, Rhineland-Palantine
  - Clinical Center "Mutterhaus" Trier, Trier, Rhineland-Palatinate
  - CaritasClinic Saarbrücken, Saarbrücken, Saarland
  - Clincal Center Chemnitz, Chemnitz, Saxony
  - Radiotherapy Practice Dr. A. Schreiber, Dresden, Dresden, Saxony
  - Oncology Practice Dresden, Dresden, Saxony
  - University Clinic Leipzig, Leipzig, Saxony
  - Clinic Sankt Georg gGmbH, Leipzig, Leipzig, Saxony
  - University Clinic Magdeburg, Magdeburg, Saxony-Anhalt
  - University Clinic Kiel, Kiel, Schleswig-Holstein
  - Vivantes Clincial Center in Friedrichshain, Berlin
  - Clincal Center Helios Berlin Buch, Berlin
  - Ev. Waldkrankenhaus, Spandau,, Berlin
  - Helios Klinikum Berlin Emil von Behring, Berlin
  - Klinikum Bielefeld, Bielefeld
  - Onkologische Schwerpunktpraxis, Darmstadt
  - Department of Radiooncology, Frankfurt
  - Praxis für Hämatologie und Onkologie, Giessen
  - Universitätsklinikum Halle, Halle
  - Alexianer Krefeld GmbH / Maria Hilf Krankenhaus, Krefeld
  - Uniklinik Schleswig Holstein, Lübeck
  - Dietrich Bonhoeffer Klinik, Neubrandenburg
  - Med. Statistik Saarbrücken GgR, Saarbrücken
  - Schwarzwald-Baar-Kliniken, Villingen-Schwenningen